CLINICAL TRIAL: NCT05739305
Title: Death Certificate Analysis and Mortality at a Hospital From Colombian Orinoquia: A Retrospective Observational Trial.
Brief Title: Death Certificate Analysis at Colombian Orinoquia: A Retrospective Observational Trial.
Status: Completed | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU Director, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2023_01
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hospital Mortality; Cancer; Chronic Disease; Non Communicable Chronic Diseases; Public Health
Keywords: Death Certificate; Hospital Mortality; Epidemiology; Public Health; Cancer; Geriatrics; Neoplasms; Colombian Orinoquia; Colombia
MeSH Terms: conditions — Neoplasms; Chronic Disease; Noncommunicable Diseases | interventions — Risk Factors; Cause of Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cancer: Death certificates of patients died by cancer or with cancer.
  Interventions: Other: Risk factor
- Cardiovascular: Death certificates of patients died by cardiovascular conditions or complications.
  Interventions: Other: Risk factor
- Tuberculosis: Death certificates of patients died by or with tuberculosis, including patients with HIV.
  Interventions: Other: Risk factor
- Infants: Death certificates of pediatric patients with more than a month of birth, and less than 18 years old.
  Interventions: Other: Risk factor
- Congenital malformations: Death certificates of patients died by congenital malformations, independently of age.
  Interventions: Other: Risk factor
- Maternal: Death certificates of patients died by obstetrical conditions during pregnancy or delivery.
  Interventions: Other: Risk factor
- Contagious: Death certificates of patients died by contagious/infectious diseases.

INTERVENTIONS:
Other: Risk factor — No diagnostic or therapeutic intervention; the characteristics of subgroups will be analyzed by the cause of death certificated in the registry.
  Other Names: Cause of death
  Groups: Cancer; Cardiovascular; Congenital malformations; Infants; Maternal; Tuberculosis

SUMMARY:
By hospital mortality, the health of a population is identified. Death certificates are a valuable tool in establishing causes of death.

The objective will be to analyze the main causes of death in hospitalized patients by population groups of interest.

A retrospective observational study will be carried out, by analyzing the death databases of the Hospital Departamental of Villavicencio from January 2012 to May 2022. The records will be exported to Excel for review and debugging. Demographic variables and causes of death will be analyzed. The categorical variables will be described in frequency and proportion; the quantitative ones will be defined in their central distribution and dispersion. For comparison, the Chi-square and Mann-Whitney test will be performed according to the characteristics of the outcome studied.

It is expected to identify the main causes of death in the groups of interest (adults, maternal, infants, fetal and non-fetal, congenital malformations) and their characteristics.

DETAILED DESCRIPTION:
Hospital mortality is a measure of the effectiveness of interventions in health, and its systematic evaluation is convenient, as an indicator of clinical management. It is considered that in internal medicine services, it can be between 6-21%, which depends on its complexity. and the population of influence.

The identification of hospital causes of death (COD) makes it possible to recognize the prevailing public health problems in the population. This information is relevant for decision-making, planning, and directing public and institutional policy. Hospital mortality is an important source of these data, in a region where most deaths occur at hospital settings. The proportion of deaths in hospitals is growing internationally and in Villavicencio, this could be the case in most cases. There are few alternatives for palliative care and end-of-life care in low and middle-income countries. Few studies analyze information from hospital institutions.

Access to death indices is free in countries such as Spain, in order to allow studies on the health of the population. Even so, there is concern about the quality of the records, from health organizations, although the uncertainty that involves establishing the COD does not necessarily conflict with the precision of metrology, according to more pragmatic thoughts.

The death certificate (CD) is the main source of data on mortality. CDs are the legal record of the causes of death and are usually made by health personnel, mainly doctors. Such information is essential to establish the priorities in health policies, of each individual institution, and in the general population. They collectively indicate the state of health of a nation.

Uncertainty about the cause of death can be a significant challenge in scenarios such as unexpected death or after a prolonged period without medical attention.

Errors in completing the information on CDs are recognized as a universal problem, which can lead to confusion in the prevalence of causes of death (COD). The use of ill-defined codes and conditions (CCMD) as COD is frequent at a universal level. Some have considered that the doctor should be socialized with the vital status and COD of their patients.

ELIGIBILITY:
Inclusion Criteria:

* Deceased people during hospitalization.
* Out-of-hospital deceased people (home) and certified by the institution

Exclusion Criteria:

* Registers of people deceased by an external (violent) cause.
* Registers of people that required certification by the Coroner's office.

Max Age: 120 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population included in the study are those included in the institutional registry of death certification after they died in the hospital or somewhere else, but had to be certified by a doctor from it for any reason.
  People who died by an external cause included in chapters XIX and XX of 10-ICD were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Number of preventable deaths | 12 years
  Deaths caused by diseases or conditions potentially preventable, according to the Holland criteria, or other authors.

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez Gutierrez, MD, Principal Investigator — ICU director
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is collected from an institutional registry of deceased people retrospectively. Even when it does not contain the personal information of participants, the database will not be shared in a repository. The trial final report will be uploaded in Mendeley Data and published in an indexed journal.

REFERENCES:
- [Result] Carvajal Y, Kottow M. [The metrology of uncertainty: a study of vital statistics from Chile and Brazil]. Cad Saude Publica. 2012 Nov;28(11):2063-75. doi: 10.1590/s0102-311x2012001100006. Spanish. PMID 23147948
- [Result] Ferorelli D, Donno F, De Giorgio G, Zotti F, Dell'Erba A. Study of determinants in deaths occurring in an Italian teaching hospital during a year. Clin Ter. 2020 May-Jun;171(3):e245-e252. doi: 10.7417/CT.2020.2222. PMID 32323714
- [Result] Morgan A, Andrew T, Guerra SMA, Luna V, Davies L, Rees JR. Provider reported challenges with completing death certificates: A focus group study demonstrating potential sources of error. PLoS One. 2022 May 20;17(5):e0268566. doi: 10.1371/journal.pone.0268566. eCollection 2022. PMID 35594279
- [Result] Ng TC, Lo WC, Ku CC, Lu TH, Lin HH. Improving the Use of Mortality Data in Public Health: A Comparison of Garbage Code Redistribution Models. Am J Public Health. 2020 Feb;110(2):222-229. doi: 10.2105/AJPH.2019.305439. Epub 2019 Dec 19. PMID 31855478
- [Result] Cirera L, Segura A. [Updated medical death documents: Medical Death Certificate and the Birth Statistics Bulletin]. Aten Primaria. 2010 Aug;42(8):431-7. doi: 10.1016/j.aprim.2009.09.029. Epub 2010 May 27. Spanish. PMID 20537431
- [Result] Cendales R, Pardo C. [Colombian death certificate quality, 2002-2006]. Rev Salud Publica (Bogota). 2011 Apr;13(2):229-38. doi: 10.1590/s0124-00642011000200005. Spanish. PMID 22030881
- [Result] Murphy SL, Xu J, Kochanek KD, Arias E. Mortality in the United States, 2017. NCHS Data Brief. 2018 Nov;(328):1-8. PMID 30500322
- [Result] Viana Alonso A, Delgado Cirerol V, de la Morena Fernandez J. [Validity of the final diagnosis in the discharge reports of deceased patients in a teaching department of internal medicine]. Rev Clin Esp. 1992 Oct;191(6):323-4. Spanish. PMID 1470725
- [Result] Armstrong D. The COVID-19 pandemic and cause of death. Sociol Health Illn. 2021 Aug;43(7):1614-1626. doi: 10.1111/1467-9566.13347. Epub 2021 Jul 13. PMID 34255866
- [Result] Sainz-Otero AM, Marin-Paz AJ, Almenara-Barrios J. The Classification of Causes of Historical Mortality (CCHM): A proposal of the study of death records. PLoS One. 2020 Apr 14;15(4):e0231311. doi: 10.1371/journal.pone.0231311. eCollection 2020. PMID 32287285
- See also: Mortality in patients hospitalized in the internal medicine service of a university hospital. An article from a local journal with a study about a university hospital mortality. — http://www.actamedicacolombiana.com/ojs/index.php/actamed/article/view/1050
- See also: Tendencias en la mortalidad de médicos generales y especialistas en Cali, Colombia. Unique article exploring the cause of death of medical doctors in Cali, Colombia. — https://revistas.unilibre.edu.co/index.php/rc_salud_ocupa/article/view/4852